CLINICAL TRIAL: NCT01097499
Title: Role of Light Emitting Diode on Implant Stability, Bone Resorption and Analgesia Post Dental Implant Placement
Brief Title: Low Level Laser (LED) Use to Increase Dental Implant Stability and Post Operative Analgesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Dr. Mahdi Ghuloom, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSH-Biolux2010
Record Dates: First submitted 2010-03-31; First posted 2010-04-01 (Estimated); Last update posted 2010-04-01 (Estimated); Status verified 2010-03

CONDITIONS: Implant; Analgesia
Keywords: Dental implant initial stability; Initial bone resorption post implant placement; Analgesia effect of LED intervention
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LED application (Active Comparator): Patients in this group will be given the LED device and will be instructed on how and when to use it. They will receive LED treatment to the surgical site preoperatively by the surgeon for 20 minutes. Then, patients in this group will apply LED at home to the surgical site postoperatively at the day of surgery and for the following 9 postoperative days.
  Interventions: Device: OsseoPulse device (Light emitting diode technology)
- No LED application (No Intervention): These patients will receive conventional dental implant treatment without the application of the LED therapy.

INTERVENTIONS:
Device: OsseoPulse device (Light emitting diode technology) — Patients in this group will be given the LED device and will be instructed on how and when to use it. They will receive LED treatment to the surgical site preoperatively by the surgeon for 20 minutes. Then, patients in this group will apply LED at home to the surgical site postoperatively at the day of surgery and for the following 9 postoperative days.
  Other Names: Device by Biolux Lic# 77929 (Approved by Health Canada)
  Arms: LED application

SUMMARY:
Study hypothesis: Low level laser (LED) will reduce initial bone resorption and improve primary stability of dental implant. It will also reduces post operative pain compared to patient without treatment

Implant osseointegration depends on many factors including biocompatibility of implant materials, design, surface, surgical access, patient conditions, biomechanical status, and lack of primary stability.

Several in vivo and in vitro studies showed the healing effect of low level laser therapy (LLLT) on bone by decreasing the initial bone resorption postoperatively and increasing the primary stability of the implant. It has also shown to have an analgesic effect intraorally when used post intraoral surgical procedures. The exact mechanism is unclear despite the fact that many hypothesis has been proposed.

In our study, our goal is to present, in a randomized standardized clinical trial, the effect of LLLT on post operative implant stability assessed by resonance frequency analysis (RFA). We will assess the subjective measures of postoperative pain using visual analog scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* 1) English speaking

Exclusion Criteria:

* 1) Systemic factors: Diabetes, systemic immune disease, smoking (non-smoking is not absolute, but preferable.)
* 2) Local factors: No immediate implants, No grafting to the site, No other implants at separate location in the mouth around the same treatment period.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-08 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Implant stability | Immediately post-op, 1, 2, 4, and 8 weeks
  Implant stability and bone quality will be assessed via RFA technology using Ostelle device (Resonance Frequency Analysis technology)

SECONDARY OUTCOMES:
Post-op analgesics | Every 3 hours the day of the surgery post-op, then every morning, and at bed time for the following 7 days
  Analgesia will be assessed using a combination of VAS and categorical scale. Patient will fill a pre-printed form with the modified VAS every 3 hours at the day of surgery, and every morning and at night for 7 days. Pt. will also reports the time and the dose of analgesics they are taking post operatively to control pain in that form. Patients will submit all the data to the surgeons at the 1-week follow-up appointment

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Clokie, DDS, FRCS, Study Director — University of Toronto/Mount Sinai Hospital
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada